CLINICAL TRIAL: NCT00002585
Title: PHASE II CLINICAL EVALUATION OF PYRAZOLOACRIDINE IN PATIENTS WITH METASTATIC BREAST CANCER
Brief Title: Pyrazoloacridine in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000063706; P30CA022453 (NIH); WSU-C-1148-93; NCI-T94-0003H
Record Dates: First submitted 1999-11-01; First posted 2004-08-11 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — NSC 366140

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: pyrazoloacridine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of pyrazoloacridine in treating women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the efficacy of pyrazoloacridine (PZA) administered by 3-hour infusion in women with metastatic breast cancer. II. Assess the qualitative and quantitative toxicities of PZA on this schedule. III. Assess the response duration and survival of patients treated with this agent.

OUTLINE: All patients receive intravenous pyrazoloacridine (PZA) every 3 weeks in the absence of progressive disease or unacceptable toxicity. Therapy continues in responding patients until 6 months after a complete response or for 1 year, whichever is shorter; stable patients receive a maximum of 4 courses. The dose is increased once for patients who experience minimal toxicity. Patients who fail PZA are encouraged to continue therapy with cyclophosphamide/doxorubicin/fluorouracil (CAF). All patients are followed for survival. Prophylactic granulocyte colony-stimulating factor is not permitted.

PROJECTED ACCRUAL: Up to 20 patients will be accrued over 7-12 months. If no more than 1 response is seen in the first 12 evaluable patients, accrual will cease.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically documented breast adenocarcinoma Clinical or radiologic evidence of metastatic disease required Histologic confirmation recommended if evidence is equivocal Bidimensionally measurable disease required, i.e.: Lesion with clearly defined margins on physical exam or radiologic evaluation with 1 diameter greater than 0.5 cm Lytic bone metastases only if measurable on bone x-ray/survey Lesion previously irradiated only if subsequent measurable progression New measurable lesion in previously irradiated field The following are not considered measurable: Unidimensionally measurable lesions Palpable nodal disease not measurable on CT Masses with margins not clearly defined Lesions with both diameters less than 0.5 cm Bone disease other than lytic bone disease Pleural effusions or ascites Disease identified by bone scan only History of bilateral breast cancer allowed No brain metastases CT required if clinically indicated No meningeal carcinomatosis Hormone receptor status: Any status

PATIENT CHARACTERISTICS: Age: Over 18 Sex: Women only Menopausal status: Not specified Performance status: Zubrod 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute granulocyte count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dL Renal: Creatinine less than 1.5 mg/dL Other: No second malignancy within 5 years except: Adequately treated nonmelanomatous skin cancer Adequately treated carcinoma in situ of the cervix Not pregnant or nursing Negative pregnancy test required of premenopausal women Appropriate contraception required of fertile women Blood/body fluid analyses to determine eligibility and physical exams for tumor measurement completed within 7 days prior to registration; imaging studies to evaluate and document measurable disease completed within 4 weeks prior to registration

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No more than 1 prior chemotherapy for metastatic disease allowed At least 4 weeks since adjuvant chemotherapy Endocrine therapy: Prior hormonal therapy allowed At least 4 weeks since hormonal therapy for patients with partial or complete response to most recent maneuver Radiotherapy: Prior radiotherapy for metastatic disease allowed At least 4 weeks since radiotherapy and recovered Surgery: Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1994-02; Primary Completion 1999-10 (Actual); Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M. LoRusso, DO, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States